CLINICAL TRIAL: NCT04267640
Title: A Phase II Double-Blind, Randomized, Placebo-Controlled Study to Assess the Efficacy and Safety of AMG0001 to Improve Ulcer Healing and Perfusion in Subjects Who Have Peripheral Ischemic Ulcers of the Lower Extremity
Brief Title: Study of AMG0001 to Improve Ulcer Healing and Perfusion in Subjects With Peripheral Ischemic Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnGes USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG-CLTI-0211
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Peripheral Artery Disease; Ischaemic Ulcer of Lower Leg Due to Atherosclerotic Disease; Chronic Limb Threatening Ischemia; Ischemic Ulcer of Foot
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AMG0001 4mg (Experimental): AMG0001 4mg + standard wound care
  Interventions: Biological: AMG0001
- AMG0001 8mg (Experimental): AMG0001 8mg + standard wound care
  Interventions: Biological: AMG0001
- Placebo (Placebo Comparator): Placebo + standard wound care
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AMG0001 — AMG0001 is a DNA Plasmid encoding hepatocyte growth factor (HGF) administered intramuscularly
  Other Names: HGF plasmid; Collategene; beperminogene perplasmid
  Arms: AMG0001 4mg; AMG0001 8mg
Biological: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of intramuscular injection of AMG0001 (hepatocyte growth factor [HGF] plasmid) to improve ulcer healing and perfusion in patients with peripheral artery disease.

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, randomized, placebo-controlled, parallel group study. Approximately 60 male or female subjects aged 18 years or older with one shallow foot ulcer and mild/moderate ischemia due to peripheral artery disease (PAD) will be randomized in a 1:1:1 ratio to one of 3 treatment groups:

* 4.0 mg AMG0001 intramuscular (IM) (n = 20)
* 8.0 mg AMG0001 IM (n = 20)
* Placebo IM (n = 20)

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of PAD and mild/moderate foot ischemia (WIFI ischemia grades 1, 2)
* A single measurable ulcer of ≥ 1 cm2 and ≤ 10 cm2 on a lower extremity without evidence of infection or gangrene and no evidence of bone and/or tendon involvement at randomization
* Subjects will undergo protocol-defined standardized wound care during the screening period and through 12 months from the first dose of investigational product
* Subjects who have a diagnosis of diabetes must be considered stable with no changes in diabetic medication regimen anticipated during the study period. Subjects who have a diagnosis of diabetes must have a HbA1c of ≤12% at Screening

Exclusion Criteria:

* Subjects who have excessive tissue necrosis that is unlikely to benefit from medication, or those subjects who, in the opinion of the Investigator, are felt likely to require revascularization within 1 month of screening
* Subjects with severe limb ischemia
* Subjects who are considered likely to require a major amputation (at or above the ankle) within 3 months of screening
* Subjects with deep ulcerations with bone or tendon exposure, or uncontrolled infection, or with the largest ulcer that is >10 cm2 in area
* Subjects with hemodynamically significant aorto-iliac occlusive disease
* Subjects who have had a technically successful revascularization by surgery or angioplasty within 2 months. If subjects are more than two months from revascularization and still meet the inclusion criteria, they may be considered for enrollment. Subjects who have had a technically unsuccessful attempt at revascularization may be enrolled at least one week from the procedure
* Subjects currently receiving immunosuppressive medication, systematically administered steroid therapy, chemotherapy or radiation therapy. Inhaled and topical steroid therapies are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Complete ulcer healing at 6 months | Month 6
  Complete ulcer healing defined as skin re-epithelialization without drainage or dressing requirements confirmed at 2 consecutive study visits 2 weeks apart.
Time to complete ulcer healing | Month 12
  Complete ulcer healing defined as skin re-epithelialization without drainage or dressing requirements confirmed at 2 consecutive study visits 2 weeks apart.

SECONDARY OUTCOMES:
The percentage reduction of ulcer size from baseline | Months 4, 6, 8, 10, 12
Hemodynamic measurements of toe pressure (TP) | Months 4, 6, 8, 10, 12
  Measure of baseline and change from baseline for hemodynamic parameters
Hemodynamic measurements of ankle systolic pressure (ASP) | Months 4, 6, 8, 10, 12
  Measure of baseline and change from baseline for hemodynamic parameters
Hemodynamic measurements of ankle brachial index (ABI) | Months 4, 6, 8, 10, 12
  Measure of baseline and change from baseline for hemodynamic parameters
Hemodynamic measurements of toe brachial index (TBI) | Months 4, 6, 8, 10, 12
  Measure of baseline and change from baseline for hemodynamic parameters
Hemodynamic measurements of TcPO2 | Months 4, 6, 8, 10, 12
  Measure of baseline and change from baseline for hemodynamic parameters
Visual Analogue Scale (VAS) | Months 4, 6, 8, 10, 12
  Measure of baseline and change from baseline for VAS. VAS is a 10-cm line (with score ranges 0 to 10), oriented horizontally; the left end of the line (0 mark) indicates "no pain"; the right end indicates "pain as bad as it can be."
Occurrence of New Ulcer of the Index leg | Months 4, 6, 8, 10, 12
  Number of subjects and proportions with new ulcer
Major / Minor Amputations (digit, forefoot) / Revascularization of the Index Leg | Months 4, 6, 8, 10, 12
  Number of subjects and proportions with major/minor amputation or revascularization

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, MD, DPM, PhD, Principal Investigator — Keck School of Medicine USC; Michael S Conte, MD, Principal Investigator — Division of Vascular and Endovascular Surgery, UCSF
Locations (20):
- United States (20):
  - ILD Research Center, Carlsbad, California
  - Rancho Research Institute, Downey, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Felix Sigal, D.P.M. A Professional Corporation, Los Angeles, California
  - Center for Clinical Research Inc., San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Goleta Valley Cottage Hospital, Santa Barbara, California
  - BRCR Global, Deerfield Beach, Florida
  - Doctors Research Network, South Miami, Florida
  - Barry University Clinical Research, Tamarac, Florida
  - Guardian Research/Florida Cardiology, Winter Park, Florida
  - Gateway Clinical Trials, LLC, Belleville, Illinois
  - Rosalind Franklin University Health Clinics, North Chicago, Illinois
  - Brigham and Women's Hospital / Harvard Medical School, Boston, Massachusetts
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Vascular Solutions of North Carolina, Cary, North Carolina
  - The Lindner Center for Research and Education at the Christ Hospital, Cincinnati, Ohio
  - Lower Extremity Institute for Research and Therapy (LEIRT), Youngstown, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Foot and Ankle Associates of Southwest Virginia, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Armstrong DG, Conte MS, Mills JL, Menard MT, Orgill DP, Galiano RD, Kirsner RS, Farber A, Lantis JC, Zelen CM, Carter MJ, Hicks CW, Powell RJ. Anatomically Directed Lower Extremity Gene Therapy for Ulcer Healing: A Double-Blind, Randomized, Placebo-Controlled Study (LEGenD-1). Circ Cardiovasc Interv. 2025 Nov 4:e015648. doi: 10.1161/CIRCINTERVENTIONS.125.015648. Online ahead of print. PMID 41186002